CLINICAL TRIAL: NCT03036865
Title: A Double-blind, Phase 1, Single Ascending Dose Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of BOS161721 in Healthy Subjects
Brief Title: Study to Assess the Safety, Pharmacokinetics and Pharmacodynamics of BOS161721 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BOS161721-01; PXL232187 (Other: PAREXEL)
Record Dates: First submitted 2017-01-27; First posted 2017-01-30 (Estimated); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Healthy Participants
Keywords: Healthy participants; BOS161721; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (15):
- Cohort 1: 1 mg, IV BOS161721 (Experimental): Each participant will receive a single intravenous (IV) dose of BOS161721 1 milligram (mg).
  Interventions: Drug: BOS161721
- Cohort 1: matching placebo (Placebo Comparator): Each participant will receive matching IV placebo.
  Interventions: Drug: Placebo
- Cohort 2: 3 mg, SC BOS161721 (Experimental): Each participant will receive a single subcutaneous (SC) dose of BOS161721 3 mg.
  Interventions: Drug: BOS161721
- Cohort 2: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo
- Cohort 3: 10 mg, SC BOS161721 (Experimental): Each participant will receive a single SC dose of BOS161721 10 mg.
  Interventions: Drug: BOS161721
- Cohort 3: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo
- Cohort 4: 30 mg, SC BOS161721 (Experimental): Each participant will receive a single SC dose of BOS161721 30 mg.
  Interventions: Drug: BOS161721
- Cohort 4: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo
- Cohort 5: 60 mg, SC BOS161721 (Experimental): Each participant will receive a single SC dose of BOS161721 60 mg.
  Interventions: Drug: BOS161721
- Cohort 5: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo
- Cohort 6: 22 mg, IV BOS161721 (Experimental): Each participant will receive a single IV dose of BOS161721 22 mg.
  Interventions: Drug: BOS161721
- Cohort 7: 120 mg, SC BOS161721 (Experimental): Each participant will receive a single SC dose of BOS161721 120 mg.
  Interventions: Drug: BOS161721
- Cohort 7: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo
- Cohort 8: 240 mg, SC BOS161721 (Experimental): Each participant will receive a single SC dose of BOS161721 240 mg.
  Interventions: Drug: BOS161721
- Cohort 8: matching placebo (Placebo Comparator): Each participant will receive matching SC placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BOS161721 — Single dose administered IV or SC
  Arms: Cohort 1: 1 mg, IV BOS161721; Cohort 2: 3 mg, SC BOS161721; Cohort 3: 10 mg, SC BOS161721; Cohort 4: 30 mg, SC BOS161721; Cohort 5: 60 mg, SC BOS161721; Cohort 6: 22 mg, IV BOS161721; Cohort 7: 120 mg, SC BOS161721; Cohort 8: 240 mg, SC BOS161721
Drug: Placebo — Single dose administered IV or SC
  Arms: Cohort 1: matching placebo; Cohort 2: matching placebo; Cohort 3: matching placebo; Cohort 4: matching placebo; Cohort 5: matching placebo; Cohort 7: matching placebo; Cohort 8: matching placebo

SUMMARY:
Study BOS161721-01 is a randomized, single center, double-blind, placebo-controlled trial conducted to study the safety, pharmacokinetics (PK), and pharmacodynamics (PD) of single ascending intravenous (IV) and subcutaneous (SC) doses of BOS161721 or placebo in healthy adult male and female participants.

DETAILED DESCRIPTION:
Study BOS161721-01 will consist of 7 single ascending dose (SAD) cohorts, each with 8 participants (6 active:2 placebo), and an eighth SAD cohort with 5 participants (all active). Participants will be randomized in a 3:1 ratio (BOS161721:placebo) and will either receive a single dose of BOS161721 (1, 3, 10, 22, 30, 60, 120, or 240 milligrams [mg]) or placebo. Participants in Cohort 1 will receive the lowest dose, administered IV (1 mg), followed by Cohort 2, in which participants will receive the second lowest dose, administered SC (3 mg). BOS161721 or placebo will also be administered SC in Cohorts 3, 4, 5, 7, and 8. Participants in Cohort 6 will be administered an IV dose of 22 mg (5 active) in parallel to the 60 mg SC-dosed fifth cohort. This dose has been selected to generate a similar exposure to that following the 30 mg SC dose. The actual Cohort 6 IV dose may be adjusted upon available PK data.

Participants will be in this study for up to 56 weeks, which includes a Screening Period of up to 28 days, a single-dose treatment day (during the in-subject treatment period), and a 52-week post-treatment Follow-up Period, which is required due to the potential half-life of BOS161721.

ELIGIBILITY:
Inclusion Criteria:

* Participant voluntarily agrees to participate in this study and signs an Institutional Review Board (IRB)-approved informed consent prior to performing any of the Screening procedures
* Participants should be between 18 and 55 years (both inclusive) of age at the time of Screening, with a body mass index (BMI) between 17.5 and 32 kilograms per meters squared (kg/m^2) (both inclusive) at the time of Screening, have a weight > 50 kg and < 120 kg at the time of Screening, and be in general good health at least 8 weeks prior to the Screening visit. Good health is defined as individuals without known disease(s) as determined by a responsible physician, based on medical evaluation, including medical history, physical examination, laboratory tests, imaging, and cardiac monitoring.
* Women of non-childbearing potential status:

  * Hysterectomy;
  * Bilateral tubal ligation/tubal occlusion;
  * Bilateral salpingectomy;
  * Bilateral oophorectomy;
  * Postmenopausal - defined as 12 months of spontaneous amenorrhea (In questionable cases, a blood sample will be taken with simultaneous testing of follicle-stimulating hormone (FSH) and estradiol levels, which should be consistent with menopausal range.)
* Women of childbearing potential will be allowed to participate and have to agree to use at least 1 of the following contraception methods at all times throughout study participation in addition to either a condom with spermicide or a diaphragm/cervical cap with spermicide:

  * Non-hormonal intrauterine device (IUD; Paragard®/copper)
  * Hormonal IUD (Mirena®)
  * Nexplanon® or implantation - progesterone inserts under the skin
* Males will either be sterile, agree to be abstinent from Day -1 through the last study visit, or agree to use 2 highly effective methods of contraception such as:

  * A male condom with spermicide;
  * A sterile sexual partner;
  * Use by female sexual partner of an IUD with spermicide; a female condom with spermicide; contraceptive sponge with spermicide; an intravaginal system; a diaphragm with spermicide; a cervical cap with spermicide; or oral, implantable, transdermal, or injectable contraceptive(s).
* Non-smokers or people who smoke up to 5 cigarettes per day but less than 10 packs per year
* Participants should be willing and able to comply with all study procedures. The criterion for inclusion will be reviewed and verified at Screening and admission.

Exclusion Criteria:

* Prior clinical trial experience with monoclonal antibodies if there were clinically relevant tolerability issues with previous administration or if a washout period of 60 days or 5 half-lives (whichever is longer) has not occurred prior to the planned first day of dosing
* History of any autoimmune disease (e.g., rheumatoid arthritis, Lupus)
* History or current diagnosis of cancer, with the exception of non-melanoma skin cancer or cervical cancer in situ treated with apparent success with curative therapy (response duration > 5 years)
* Asthma, currently treated with or in the opinion of the Principal Investigator likely to require additional systemic glucocorticosteroid therapy during the study, is exclusionary.
* History of any clinically important drug or vaccine allergy or anaphylaxis
* A cluster of differentiation 4 (CD4+) lymphocyte count < 500 cell/millimeters cubed (mm^3) at Screening
* Positive anti-keyhole limpet hemocyanin (KLH) antibodies at Screening
* Previous immunization with KLH
* Known allergy to shellfish, KLH vaccine, or hypersensitivity to proteins foreign to the body
* Levels of Immunoglobulin G (IgG) and Immunoglobulin M (IgM) outside of reference value deemed clinically significant by the Principal Investigator at Screening
* History or sensitivity to heparin or heparin-induced thrombocytopenia
* Participants with cryptosporidium in the stool sample at Screening
* Abnormal bilirubin or alanine aminotransferase (ALT) at Screening as judged by the Principal Investigator to be clinically significant
* Positive urine drug screen at Screening or Day -1
* History of alcohol dependence as determined by a positive alcohol serum test at Screening or Day -1 or participants who consume more than 14 (female participants) or 21 (male participants) units of alcohol a week (unit = 1 glass of wine [125 milliliters (mL)/4 ounces] = 1 measure [25 mL/1 ounce] of spirits = 284 mL [10 ounces] of beer)
* Participants who have a positive test, or have been treated, for Hepatitis A, Hepatitis B, Hepatitis C virus, human immunodeficiency virus (HIV), cytomegalovirus (CMV) or Epstein-Barr virus (EBV). Regarding Hepatitis B, any of the following would exclude the participant from the study:

  * Participants with positive Hepatitis B Surface antigen (HBsAg);
  * Participants with Hepatitis B DNA levels > 200 copies/mL (quantified by real-time polymerase chain reaction) in case the participant is positive for Hepatitis B surface antibody (HBsAb) but negative for HBsAg;
  * Positive for Hepatitis B core antibody (HBcAb)
* Current clinical, radiographic, or laboratory evidence of active tuberculosis (TB)
* A history of active TB within the last 3 years before Screening, even if treated
* Therapy for latent TB that has not been completed as per local country guidelines
* Positive interferon gamma release assay (IGRA) for TB unless proper treatment is documented, as described above
* Donation of blood (> 500 mL) or blood products within 2 months (56 days) prior to Day -1
* Any medically relevant pre-existing condition that could jeopardize the safety of the participant during the trial
* Any participant, on the judgment of the Principal Investigator, who would be considered unsuitable for the clinical trial
* A shingles infection in the last 6 months prior to Screening
* Live vaccination or use of steroids in the last 2 months prior to Screening
* Use of prescription medications (except for oral contraceptive) and over-the-counter treatments, including herbal supplements such as St. John's Wart (except multivitamins), in the 2 weeks prior to Screening
* Participants with poor dental health and/or severe foot fungal infections, as judged by the Principal Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01; Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Number of participants with any treatment-emergent serious adverse event (TESAE) | up to 52 weeks
Number of participants with any treatment-emergent non-serious adverse event (TEAE) | up to 52 weeks
Number of participants with TESAEs of the indicated severity | up to 52 weeks
Number of participants with TEAEs of the indicated severity | up to 52 weeks
Number of participants with abnormal, clinically significant electrocardiogram findings | Days -1 and 4 (Residential Period); Days 15, 30, and 90 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Number of participants with abnormal, clinically significant vital sign (blood pressure, heart rate, temperature) values | Screening; Days -1, 1, 2, 4, and 7 (Residential Period); Days 15, 30, 44, 60, 90, 180, 210, 270, and 360 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Number of participants with abnormal, clinically significant hematology parameter values | Screening; Days -1, 1, 2, 4, and 7 (Residential Period); Days 15, 30, 44, 60, 90, 180, 210, 270, and 360 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Number of participants with abnormal, clinically significant clinical chemistry parameter values | Screening; Days -1, 1, 2, 4, and 7 (Residential Period); Days 15, 30, 44, 60, 90, 180, 210, 270, and 360 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Mean total immunoglobulin G (IgG) levels | Screening; Days -1 and 4 (Residential Period); Days 15, 30, 60, 210 and 270 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Mean total immunoglobulin M (IgM) levels | Screening; Days -1 and 4 (Residential Period); Days 15, 30, 60, 210 and 270 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Mean cluster of differentiation 4 (CD4+) cell count | Screening; Days -1, 4, and 7 (Residential Period); Days 15, 30, 44, 60, 90, 180, 210, 270, and 360 (Follow-up Period)
  Single-day dosing will occur on Day 1.
Number of participants with abnormal, clinically significant physical examination findings | Screening; Day -1 (Residential Period)
  Single-day dosing will occur on Day 1.
Number of participants with abnormal, clinically significant targeted physical examination findings | Day 7 (Residential Period); Days 15, 44, 90, 180, 270, and 360 (Follow-up Period)
  Single-day dosing will occur on Day 1.

SECONDARY OUTCOMES:
Mean maximum observed concentration (Cmax) of intravenous (IV) BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean Cmax of subcutaneous (SC) BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Mean first time to maximum concentration (Tmax) of IV BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean Tmax of SC BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Mean area under the concentration-time curve (AUC) of IV BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean AUC of SC BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Mean terminal elimination half-life (t½) of IV BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean t½ of SC BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Mean systematic clearance (CL) of IV BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean CL of SC BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Mean volume of distribution (Vd) of IV BOS161721 | Day 1 of Cohorts 1 and 6: predose, at the end of infusion/injection (30 minutes); at 0.5, 1, 2, 4, 8, and 12 hours postdose. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 1 and 6.
Mean Vd of SC BOS161721 | Day 1 of Cohorts 2, 3, 4, 5, 7, and 8: predose; following subcutaneous injection on Day 1. Postdose on Days 2, 4, 7, 15, 30, 44, 90, 180, 210, 270, and 360 for Cohorts 2, 3, 4, 5, 7, and 8.
Number of participants with anti-drug antibodies (ADA) to BOS161721 | up to Day 60

CONTACTS AND LOCATIONS:
Locations (1):
- Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hussaini A, Mukherjee R, Berdieva DM, Glogowski C, Mountfield R, Ho PTC. A Double-Blind, Phase I, Single Ascending Dose Study to Assess the Safety, Pharmacokinetics, and Pharmacodynamics of BOS161721 in Healthy Subjects. Clin Transl Sci. 2020 Mar;13(2):337-344. doi: 10.1111/cts.12715. Epub 2019 Nov 29. PMID 31664766